CLINICAL TRIAL: NCT06889844
Title: Observational Cross-reactivity Study to Evaluate the Specificity of a Blood Test for Colorectal Cancer Diagnosis Based on Molecular Markers and Risk Factors Identified With Artificial Intelligence Tools
Brief Title: Observational Cross-reactivity Study for Colorectal Cancer Diagnosis
Status: Recruiting | Type: Observational
Sponsor: ADVANCED MARKER DISCOVERY S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMD-CCR-2022-01
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer or Gastrointestinal Disease: A different types of cancer and gastrointestinal disease will be included in the cohort such as breast cancer, bladder cancer, IBDs, Leukemia and Lung cancer.
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Patients will donate a blood sample for molecular analysis of molecular biomarkers in plasma, which being the only procedure in the study.

SUMMARY:
The objective of this observational study is to evaluate the false positive rate of the blood test based on molecular biomarkers and risk factors. A total of 250 patients diagnosed with various cancers and gastrointestinal diseases will be enrolled. The main question to be answered is

Does the blood test have a low false positive rate in the main study population?

Participants will donate a blood sample as part of their regular medical care for cancer diagnosis and give the consent to know their clinical risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age at the time of blood sample collection.
* Subjects must be able to understand the information provided on the participant information sheet, must consent to participate in the study, and must sign the informed consent form.
* Patients diagnosed with only one type of cancer (no colorectal cacner) or gastrointestinal disease.

Exclusion Criteria:

* Patients who have received previous chemotherapy or radiotherapy.
* In case of diagnosis of a tumor: patients who have undergone total or partial surgical resection of the tumor.
* Patients with a personal history of advanced or non-advanced colorectal adenoma, serrated lesions, colorectal cancer, familial adenomatous polyposis or Lynch syndrome.
* Patients without appropriate staging or diagnosis.
* Patients with hemolyzed plasma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled with a only one diagnosis of cancer (no colorectal cancer) or gastrointestinal disease at the time of a consultation within the Oncology, Digestive System, Gastroenterology, Endoscopy or Surgery Service. Patients will be included in a competitive, consecutive and progressive manner by the Centers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
False Positive Rate | 36 month
  To estimate the false positive rate of the blood-based test in the main population of the study

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospitales HM de Malaga, Málaga, Andalusia
  - Hospital Centro Médico Asturias, Oviedo, Cantabria
  - Hospital Universitario de Ourense, Ourense, Galicia
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - MD Anderson Cancer Centre, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579
- [Background] Herreros-Villanueva M, Duran-Sanchon S, Martin AC, Perez-Palacios R, Vila-Navarro E, Marcuello M, Diaz-Centeno M, Cubiella J, Diez MS, Bujanda L, Lanas A, Jover R, Hernandez V, Quintero E, Jose Lozano J, Garcia-Cougil M, Martinez-Arranz I, Castells A, Gironella M, Arroyo R. Plasma MicroRNA Signature Validation for Early Detection of Colorectal Cancer. Clin Transl Gastroenterol. 2019 Jan;10(1):e00003. doi: 10.14309/ctg.0000000000000003. PMID 30702491
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338